CLINICAL TRIAL: NCT03974165
Title: Functional Cereal-based Products Fortified With Legumes for Satiety and Weight Management
Brief Title: Cereal-based Products Fortified With Legumes and Effects on Glycemic Control and Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Research and Teaching Associate-Staff, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 923.20-3-2019
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-06

CONDITIONS: Appetite
Keywords: cereal-based products fortified with legumes; appetite regulation; postprandial glucose response; postprandial hormone responses

STUDY DESIGN:
Intervention Model Description: 1. Healthy subjects with normal body weight receive different cereal-based products fortified with legumes or reference food in a randomized crossover design. Postprandial glycemic and hormonal responses are evaluated.
  2. Overweight subjects receive different cereal-based products fortified with legumes or reference food in a randomized crossover design. Postprandial glycemic and hormonal responses are evaluated.
Who Masked: Participant
Masking Description: Foods do not differ in shape or color. Participants are blinded to the treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cereal-legume product 1 (Experimental): Treatment with cereal-legume product-1
  Interventions: Other: Cereal-legume product 1
- Cereal-legume product 2 (Experimental): Treatment with cereal-legume product-2
  Interventions: Other: Cereal-legume product 2
- Cereal product (Experimental): Treatment with cereal product
  Interventions: Other: Cereal product
- Reference food (Active Comparator): Treatment with reference food
  Interventions: Other: Reference food

INTERVENTIONS:
Other: Cereal-legume product 1 — The intervention examines the effect of cereal based product fortified with legumes-1 in appetite regulation in 1) subjects with normal body weight and 2) overweight subjects.
  Arms: Cereal-legume product 1
Other: Cereal-legume product 2 — The intervention examines the effect of cereal based product fortified with legumes-2 in appetite regulation in 1) subjects with normal body weight and 2) overweight subjects.
  Arms: Cereal-legume product 2
Other: Cereal product — The intervention examines the effect of cereal product in appetite regulation in 1) subjects with normal body weight and 2) overweight subjects.
  Arms: Cereal product
Other: Reference food — The intervention examines the effect of reference food in appetite regulation in 1) subjects with normal body weight and 2) overweight subjects.
  Arms: Reference food

SUMMARY:
Legumes are rich source of proteins and dietary fibers which are associated with satiety and amelioration of postprandial glycemic response. The purpose of the study is to examine the effects of cereal-based products fortified with legumes on appetite regulation and body weight management.

DETAILED DESCRIPTION:
Postprandial glycemic response as well as response of hormones related to appetite regulation after consumption of cereal-based products fortified with legumes will be evaluated. Apparently healthy subjects with normal body weight and overweight subjects will participate in the study (two protocols). Certain effects on metabolites related to the composition of the different products will be examined. The results of the study will help in the design of a long-term clinical trial regarding the effects of the functional products on body weight management in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* normal exercise and dietary habits
* weight stable for at least 3 months before enrollment

Exclusion Criteria:

* pregnancy
* diabetes
* chronic medical illness
* use of nutritional supplements
* regular intense exercise
* alcohol consumption >2 drinks per day

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose AUC | Time points: 0 (before food consumption), 30, 60, 90,120,180 minutes postprandially for each food (totally four times)
  Change in glucose AUC after consumption of the products compared to the AUC after consumption of the reference food

CONTACTS AND LOCATIONS:
Overall Officials: Vaios Karathanos, Study Chair — Harokopio University, School of Health Sciences and Education; Alexander Kokkinos, Principal Investigator — National and Kapodistrian University of Athens, School of Medicine; Amalia Yanni, Principal Investigator — Harokopio University, School of Health Sciences and Education
Locations (1):
- Laiko General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No